CLINICAL TRIAL: NCT04498598
Title: Structural Modification In Supraglottic Airway Device Enhances Exchange Between Supraglottic & Endotracheal Ventilation Modes
Brief Title: Structural Modification In Supraglottic Airway Device
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 20-163
Record Dates: First submitted 2020-07-13; First posted 2020-08-04 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Airway Complication of Anesthesia; Ventilation Therapy; Complications; Hypoxia; Hypoventilation
Keywords: Airway Management; Oxygenation and Ventilation; Airway Devices; Supraglottic Airway
MeSH Terms: conditions — Hypoxia; Hypoventilation; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- A/Z Airway (Experimental): Patients under general anesthesia for surgical procedures who need airway management for ventilation.
  Interventions: Device: A/Z Supraglottic airway

INTERVENTIONS:
Device: A/Z Supraglottic airway — Patient receive supraglottic airway for general anesthesia which can be converted to endotracheal ventilation reversibly

SUMMARY:
The proposed A/Z modification of a supraglottic airway (SGA) incorporates an opening in the SGA body that enables access to the endotracheal tube (ETT) through the body of the SGA without the need of using an exchange catheter, thus enabling an ETT to move in the body of the SGA and convert a supraglottic to endotracheal ventilation. In its original form an adaptor made from same material currently used in the endotracheal tubes can make ventilation through the proposed airway device possible in exactly the same manner of a conventional SGA currently used. This adapter also known as the R-piece can be replaced with an ETT. The modification also allows placement of SGA over an existing ETT to convert and endotracheal (ET) to supraglottic (SG) mode of ventilation without the need to use an exchange catheter.

DETAILED DESCRIPTION:
The special design allows conversion of a telescopic coaxial portion (R piece), replacing with an ETT which can act coaxially to provide both supraglottic (up position) and endotracheal (down position) of ETT. See this modification in https://www.youtube.com/watch?v=iy84lALU1aI

Currently the proposed change to the conventional SGA has been made and feasibility tested on Manikins. The A/Z airway modification is also demonstrated in the attached link video https://www.youtube.com/watch?v=ukLOAC55iG8

In this study, we are trialing the A/Z concept on an original A/Z modification by a manufacturer on their currently used SGA. Thus instead of investigators making the changes by cutting a channel in a conventional SGA immediately before use in the Operating Room, they have asked a manufacturer to do so professionally.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients
2. scheduled for a general anesthesia procedure with ETT & muscle relaxation

Exclusion Criteria:

1. Patients who are not able to consent
2. Non English Speaking
3. History of difficult airway
4. Physical exam of airway which suggests difficulty in airway management or need to use special equipment
5. BMI >35
6. Gastroesophageal reflux disease
7. Anesthetic plan other than general anesthesia
8. Emergency procedures

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Test effect of A/Z modification of supraglottic airway device on rate of successful oxygenation and ventilation before beginning a full clinical trial | During and immediately after the intervention
  An alteration and structural modification in the supraglottic airway device can improve safety of airway exchange in patient needing general anesthesia, this proof of concept should show if the modification has any affect on oxygenation and ventilation.

SECONDARY OUTCOMES:
Rate of successful exchange from supraglottic to endotracheal ventilation using A/Z modified SGA | During and immediately after intervention
  Evaluate if a modification of configuration on "Laryngeal Mask Airway" improves safety during Supraglottic to Endotracheal conversion without using an exchange catheter
Rate of successful exchange from endotracheal to supraglottic ventilation using A/Z modified SGA | During and immediately after intervention
  Evaluate if this modification can enhance smooth extubation after endotracheal intubation by converting an endotracheal tube to a supraglottic airway

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Journal Abstracts — https://doi.org/10.1093/bja/aex194 — A. Varvinskiy, T. Hinde, 21st Annual Scientific Meeting of the Difficult Airway Society: lessons learned and glimpses of the future , BJA: British Journal of Anaesthesia, Volume 119, Issue 3, September 2017, Pages e31-e47,
- Available data/document: Journal Abstacts — https://doi.org/10.1016/j.bja.2018.02.037 — J. Law, I. Morris, Historical cohort study of 10 288 tracheal intubations facilitated by video laryngoscopy, British Journal of Anaesthesia, Volume 121, Issue 1, 2018, Pages e1-e2, ISSN 0007-0912, https://doi.org/10.1016/j.bja.2018.02.037. (https://www.sciencedirect.com/science/article/pii/S0007091218301831)